CLINICAL TRIAL: NCT07342699
Title: Microsurgical Outcomes and Prognostic Analysis of 450 Cases of Cerebellar Gliomas: Integrating Pathology, Molecular Biomarkers, and Novel Clinical Insights
Brief Title: Location-Molecular Integrated Outcomes in 450 Cerebellar Glioma Microsurgical Cases
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Other Study IDs: WestChinaH-HX-2025-09
Record Dates: First submitted 2025-12-25; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2024-12

CONDITIONS: Gliomas
Keywords: Microsurgery; Prognostic factor; Molecular biomarker; Survival analysis
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cerebellar hemisphere: Tumors arise from Cerebellar hemisphere
- Vermis: Tumors arise from Cerebellar Vermis
- Fourth ventricle: Tumors arise from Fourth ventricle
- Pontocerebellar-angle (PCA) region: tumors from Pontocerebellar-angle (PCA) region

SUMMARY:
The goal of this observational study is to learn if refined anatomical location-combined with molecular biomarkers-can predict surgical success and long-term survival in 450 adults and children with cerebellar gliomas who underwent microsurgical resection at a single center between 2014 and 2024. The main questions it aims to answer are:

1. Does tumor location (cerebellar hemisphere, vermis, fourth ventricle, or pontocerebellar-angle region) independently influence extent of resection and overall survival after adjustment for WHO grade and molecular profile?
2. Among IDH-wild-type low-grade gliomas, does gross-total resection plus early adjuvant radiotherapy improve 5-year overall and progression-free survival compared with lesser resection or radiotherapy omission?

Researchers compared four anatomical subgroups and multiple molecular subtypes (IDH, 1p/19q, MGMT, TERT, BRAF V600E) to quantify location-specific resection rates, complication rates, and survival outcomes. Participants underwent standardized pre-operative imaging, microsurgical resection with intra-operative monitoring when indicated, post-operative MRI within 48 h to quantify residual tumor, and longitudinal clinical and radiographic follow-up every 3-12 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria

* Pathologically proven cerebellar glioma (hemisphere, vermis, fourth ventricle, or pontocerebellar-angle region) per 2021 WHO CNS classification
* First microsurgical resection performed at our center between January 2014 and January 2024
* Age ≥ 3 years at surgery
* Pre-operative Karnofsky Performance Status (KPS) recorded
* Availability of post-operative contrast MRI for resection-extent calculation
* Minimum required molecular data: IDH1/2 status (immunohistochemistry ± sequencing)
* Continuous follow-up ≥ 6 months after surgery (out-patient visits or telephone confirmation)

Exclusion Criteria

* Brain-stem glioma with secondary cerebellar invasion
* Recurrent or metastatic glioma
* Previous cranial radiation or glioma surgery at another institution
* Palliative resection (< 20 % of tumor volume removed)
* Missing post-operative MRI or insufficient tissue for mandatory IDH testing
* Follow-up < 6 months or lost to follow-up before 6-month landmark

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population Description The study group is 450 consecutive patients treated at a single high-volume neuro-oncology center (West China Hospital and its Longquan branch) who underwent primary microsurgical resection for a newly diagnosed glioma that arose wholly within the cerebellum.
  * **Age span**: 3-78 years (median 38 years); 52.7 % ≤ 40 y, 47.3 % > 40 y
  * **Sex**: 244 males (54.3 %), 206 females (45.7 %)
  * **Tumor origin by cerebellar sub-site**
  * Cerebellar hemisphere 223 (49.6 %)
  * Vermis 141 (31.3 %)
  * Fourth ventricle 67 (14.9 %)
  * Pontocerebellar-angle region 19 (4.2 %)
  * **WHO grade at resection**: Low-grade (I-II) 291 (64.7 %); High-grade (III-IV) 159 (35.3 %)
  * **Pre-operative functional status**: Median KPS 80 (IQR 70-90)
  * **Molecular profile (full cohort tested)**
  * IDH-mutant 152 (33.7 %), IDH-wild-type 298 (66.3 %)
  * 1p/19q codeleted 97 (21.5 %)
  * MGMT promoter methylated 161 (35.7 %)
  * TERT promoter mutant 83 (18.4 %)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) time | 6 months
  the number of months from the date of microsurgical resection to the date of death from any cause or last confirmed follow-up, measured for all 450 enrolled patients and compared across the four anatomical cerebellar locations and the predefined molecular sub-groups.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  Time from surgery (or diagnosis) to radiographic or clinical tumor progression. Used to assess efficacy of resection and adjuvant therapies.
Extent of Resection (EOR) | 6 months
  Categorized as:
  Gross Total Resection (GTR; ≥95% tumor removal) Subtotal Resection (STR; <95%) Biopsy only Correlated with survival and recurrence risk.
Rate of Postoperative Complications | 6 months
  Examples:
  Cerebellar mutism syndrome Wound infection / CSF leak Hematoma requiring reoperation Pseudomeningocele Need for ventriculoperitoneal (VP) shunt

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol